CLINICAL TRIAL: NCT03319251
Title: Biomarkers of Clinical Responsiveness to Photodynamic Therapy
Brief Title: Biomarker Database Registry for Photodynamic Therapy
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Edward Maytin, MD, PhD, Physician, The Cleveland Clinic
Other Study IDs: 16-1615
Record Dates: First submitted 2017-10-12; First posted 2017-10-24 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood samples will be collected on the date of Photodynamic Therapy. A total of 13.5mL of blood will be collected between 2 tubes (3.5mL gold top tube and a 10 mL lavendar top Vacutainer tube with EDTA). The biomarkers to be examined include serum VitD levels at the time of PDT, and the presence/absence of gene alleles that correlate with expression of several proteins involved in VitD and 5FU metabolism.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research is to obtain a blood sample from patients with actinic keratoses undergoing routine Photodynamic Therapy, in order to measure biomarkers that are relevant to VitD and 5FU metabolism and might be predictive of PDT outcome. The biomarkers to be examined include serum VitD levels at the time of PDT, and the presence/absence of gene alleles that correlate with expression of several proteins involved in VitD and 5FU metabolism. The presence of these biomarkers will be correlated to the improvement in AK lesion counts at the patient's routine follow-up visit 3 months after PDT treatment.

DETAILED DESCRIPTION:
Patients who have been scheduled to receive PDT in our noninvasive cutaneous oncology clinics will be given written information prior to their visit, including a copy of the Informed Consent (IC) that describes the purpose of the study. If the patient indicates that he/she is interested, the physician or study nurse will review the IC with the patient on the day of PDT and answer all questions. After the patient signs the IC, the patient will have their blood drawn by a caregiver who has completed PTS Phlebotomy Training.

DNA samples will be stored in a locked minus 80 degree ultrafreezer, in Dr. Maytin's laboratory (room ND4-25A in the Lerner Research Institute). The samples will be maintained for up to 10 years.

Blood sample tubes and data sheets in the laboratory will be labeled with a code consisting of the first 5 digits of the patient's 8-digit MRN along with the date that the phlebotomy was performed (i.e. the date of the blood draw). This should ensure anonymity of the data while preventing mistakes when linking the laboratory results to the correct patient. Study personnel with password-protected access to the database registry will use the code to unequivocally identify the subject's file within the Oracle database and thereby enter the subject's laboratory results into the proper data field.

The Informed Consent document informs the subject that he/she can withdraw permission for use of their samples at any time, and explains how to do this by contacting the Principal Investigator (PI) in writing.

Information will not be disclosed to third party outside of Cleveland Clinic for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, at least 18 years of age
* Patient has nonhypertrophic actinic keratosis, at least 10 AK lesions present on the face, scalp, forearms, chest, or legs at the time of PDT treatment

Exclusion Criteria:

* taking doxycline, a photosensitizer
* using topical retinoids, since these can exacerbate the post-PDT erythema reaction
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The desired population for this study is 100 patients who have at least 10 nonhypertrophic actinic keratosis lesions present on the face, scalp, forearms, chest, or legs and are scheduled to receive Photodynamic Therapy (PDT) at the Cleveland Clinic noninvasive cutaneous oncology clinic.
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Actinic Keratosis (AK) clearance | at 3 months post-treatment
  Change in AK lesions present at 3 months post-PDT treatment
Vitamin D levels | At baseline, which is the day of PDT treatment
  Vitamin D level (25-hydroxy-cholecalciferol) measured in serum

SECONDARY OUTCOMES:
Allele polymorphisms in the gene of the Vitamin D receptor (VDR) | At baseline, which is the day of PDT treatment
  Identify the allele combination present at VDR locus
Allele polymorphisms in the gene promoter of thymidylate synthase (TS) enzyme | At baseline, which is the day of PDT treatment
  Identify the allele combination present at TS locus

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data, needs HIPPA clearance and specific IRB approval, we did not plan on original data being shared

REFERENCES:
- [Derived] Heusinkveld LE, Bullock TA, Negrey J, Warren CB, Maytin EV. Sandpaper curettage: A simple method to improve PDT outcomes for actinic keratosis. Photodiagnosis Photodyn Ther. 2022 Dec;40:103050. doi: 10.1016/j.pdpdt.2022.103050. Epub 2022 Aug 3. PMID 35932960
- [Derived] Bullock TA, Negrey J, Hu B, Warren CB, Hasan T, Maytin EV. Significant improvement of facial actinic keratoses after blue light photodynamic therapy with oral vitamin D pretreatment: An interventional cohort-controlled trial. J Am Acad Dermatol. 2022 Jul;87(1):80-86. doi: 10.1016/j.jaad.2022.02.067. Epub 2022 Mar 18. PMID 35314199